CLINICAL TRIAL: NCT04513925
Title: A Phase III, Open-Label, Randomized Study of Atezolizumab and Tiragolumab Compared With Durvalumab in Patients With Locally Advanced, Unresectable Stage III Non-Small Cell Lung Cancer Who Have Not Progressed After Concurrent Platinum-Based Chemoradiation
Brief Title: A Study of Atezolizumab and Tiragolumab Compared With Durvalumab in Participants With Locally Advanced, Unresectable Stage III Non-Small Cell Lung Cancer (NSCLC)
Acronym: SKYSCRAPER-03
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO41854; 2019-004773-29 (EudraCT Number)
Record Dates: First submitted 2020-08-13; First posted 2020-08-14 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab; Tiragolumab; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Atezolizumab + Tiragolumab (Experimental): Participants will receive atezolizumab administered intravenously (IV) on Day 1 of each 28-day cycle followed by tiragolumab administered IV on Day 1 of each 28-day cycle for a maximum of 13 cycles.
  Interventions: Drug: Atezolizumab; Drug: Tiragolumab
- Durvalumab (Active Comparator): Participants will receive durvalumab administered IV during each 28-day cycle for a maximum of 13 cycles.
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab 1680 mg every 4 weeks (Q4W) will be administered IV on Day 1 of each 28-day cycle.
  Other Names: Tecentriq; RO5541267
  Arms: Atezolizumab + Tiragolumab
Drug: Tiragolumab — Tiragolumab 840 mg Q4W will be administered IV on Day 1 of each 28-day cycle.
  Other Names: MTIG7192A; RO7092284
  Arms: Atezolizumab + Tiragolumab
Drug: Durvalumab — Durvalumab will be administered based on weight at 10 mg/kg IV every 2 weeks (Q2W) on Days 1 and 15 of each 28-day cycle, or will be administered at a fixed dose of 1500 mg IV every 4 weeks (Q4W) (for participants whose weight >/= 30 kg) on Day 1 of each 28-day cycle.
  Arms: Durvalumab

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of atezolizumab in combination with tiragolumab compared with durvalumab in participants with locally advanced, unresectable Stage III non-small cell lung cancer (NSCLC) who have received at least two cycles of concurrent platinum-based chemoradiotherapy (CRT) and have not had radiographic disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Histologically or cytologically documented NSCLC with locally advanced, unresectable Stage III NSCLC of either squamous or non-squamous histology
* Whole-body Positron Emission Tomography-Computed Tomography (PET-CT) scan, performed prior and within 42 days of the first dose of concurrent chemoradiotherapy (cCRT)
* At least two prior cycles of platinum-based chemotherapy administered concurrently with radiotherapy (RT), which must be completed within 1 to 42 days prior to randomization in the study (one cycle of cCRT is defined as 21 or 28 days)
* The radiotherapy (RT) component in the cCRT must have been at a total dose of radiation of 60 (±10 percent [%]) gray (Gy) (54 Gy to 66 Gy) administered by intensity modulated RT (preferred) or 3D-conforming technique
* No progression during or following concurrent platinum-based CRT
* A known PD-L1 result
* Life expectancy >/= 12 weeks
* Adequate hematologic and end-organ function
* Female participants must be willing to avoid pregnancy for 90 days after the final dose of tiragolumab and 5 months after the final dose of atezolizumab, or for 3 months after the final dose of durvalumab
* Male participants must remain abstinent or use a condom during the treatment period and for 90 days after the final dose of tiragolumab
* Male participants must not donate sperm during the treatment period and for 90 days after the final dose of tiragolumab

Exclusion Criteria:

* Any history of prior NSCLC and/or any history of prior treatment for NSCLC (participants must be newly diagnosed with unresectable Stage III disease)
* NSCLC known to have a mutation in the epidermal growth factor receptor (EGFR) gene or an anaplastic lymphoma kinase (ALK) fusion oncogene
* Any evidence of Stage IV disease
* Treatment with sequential CRT for locally advanced NSCLC
* Participants with locally advanced NSCLC who have progressed during or after the definitive cCRT prior to randomization
* Any Grade >2 unresolved toxicity from previous CRT
* Grade >= 2 pneumonitis from prior CRT
* Active or history of autoimmune disease or immune deficiency
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis or evidence of active pneumonitis
* History of malignancy other than NSCLC within 5 years prior to screening with the exception of malignancies with a negligible risk of metastasis or death
* Prior allogeneic stem cell or solid organ transplantation
* Active Epstein-Barr virus (EBV) infection or known or suspected chronic active EBV infection at screening
* Treatment with investigational therapy within 28 days prior to initiation of study treatment
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-cytotoxic T lymphocyte-associated protein 4, anti-T-cell immunoreceptor with Ig and ITIM domains (anti-TIGIT), anti-PD-1 and anti-PD-L1
* Any prior Grade >/= 3 immune-mediated adverse event or any unresolved Grade > 1 immune-mediated adverse event while receiving any previous immunotherapy agent other than immune checkpoint blockade agents
* Treatment with systemic immunosuppressive medication
* Women who are pregnant, or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 829 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Independent Review Facility (IRF)-assessed Progression Free Survival (PFS) in the PD-L1-positive Analysis Set (PPAS) | From randomization to the first occurrence of disease progression or death from any cause, whichever occurs first (up to approximately 114 months)
IRF-assessed PFS in the Full Analysis Set (FAS) | From randomization to the first occurrence of disease progression or death from any cause, whichever occurs first (up to approximately 114 months)

SECONDARY OUTCOMES:
Overall Survival (OS) in the PPAS | From randomization to death from any cause (up to approximately 114 months)
Investigator-assessed PFS in the PPAS | Time from randomization to the first occurrence of disease progression or death from any cause, whichever occurs first first (up to approximately 114 months)
IRF-assessed Confirmed Objective Response Rate (ORR) in the PPAS | From randomization up to approximately 114 months
Investigator-assessed Confirmed ORR in the PPAS | From randomization up to approximately 114 months
IRF-assessed Duration of Response (DOR) in the PPAS | From first occurrence of a documented objective response to disease progression or death from any cause, whichever occurs first (up to approximately 114 months)
Investigator-assessed DOR in the PPAS | From first occurrence of a documented objective response to disease progression or death from any cause, whichever occurs first (up to approximately 114 months)
Time to Confirmed Deterioration (TTCD) Assessed Using European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core (QLQ-C30) Score in the PPAS | Up to approximately 114 months
  TTCD using EORTC QLQ-C30 is an initial 10-point decrease in global health status (GHS) and physical functioning from baseline that must be held for all subsequent assessment timepoints or followed by death attributable to cancer progression. EORTC QLQ-C30: a self-reported measure, consisting of 30 questions that assess 5 aspects of participants functioning (physical, emotional, role, cognitive and social), 3 symptom scales (fatigue, nausea and vomiting and pain), GHS and quality of life (QoL), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea and financial difficulties) with a recall period of the previous week. Functioning items are scored on a 4-point scale: 1=Not at all to 4=Very much, with higher score indicating worse outcome. Symptom items (GHS and QoL) are scored on a 7-point scale: 1=Very poor to 7=Excellent. Scores will be linearly transformed with a minimum score of 0 and maximum score of 100. Higher score indicates better outcome.
OS in the FAS | From randomization to death from any cause (up to approximately 114 months)
Investigator-assessed PFS in the FAS | Time from randomization to the first occurrence of disease progression or death from any cause, whichever occurs first first (up to approximately 114 months)
IRF-assessed Confirmed ORR in the FAS | From randomization up to approximately 114 months
Investigator-assessed Confirmed ORR in the FAS | From randomization up to approximately 114 months
IRF-assessed DOR in the FAS | From first occurrence of a documented objective response to disease progression or death from any cause, whichever occurs first (up to approximately 114 months)
Investigator-assessed DOR in the FAS | From first occurrence of a documented objective response to disease progression or death from any cause, whichever occurs first (up to approximately 114 months)
TTCD Assessed Using EORTC QLQ-C30 Score in the FAS | Up to approximately 114 months
  TTCD using EORTC QLQ-C30 is an initial 10-point decrease in global health status (GHS) and physical functioning from baseline that must be held for all subsequent assessment timepoints or followed by death attributable to cancer progression. EORTC QLQ-C30: a self-reported measure, consisting of 30 questions that assess 5 aspects of participants functioning (physical, emotional, role, cognitive and social), 3 symptom scales (fatigue, nausea and vomiting and pain), GHS and quality of life (QoL), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea and financial difficulties) with a recall period of the previous week. Functioning items are scored on a 4-point scale: 1=Not at all to 4=Very much, with higher score indicating worse outcome. Symptom items (GHS and QoL) are scored on a 7-point scale: 1=Very poor to 7=Excellent. Scores will be linearly transformed with a minimum score of 0 and maximum score of 100. Higher score indicates better outcome.
IRF-assessed PFS Rates at 12 Months, 18 Months and 24 Months in the PPAS | 12, 18 and 24 months
IRF-assessed PFS Rates at 12 Months, 18 Months and 24 Months in the FAS | 12, 18 and 24 months
Investigator-assessed PFS Rates at 12 Months, 18 Months and 24 Months in the PPAS | 12, 18 and 24 months
Investigator-assessed PFS Rates at 12 Months, 18 Months and 24 Months in the FAS | 12, 18 and 24 months
OS Rates at 12 Months, 24 Months, 36 Months and 48 Months in the PPAS | 12, 24, 36 and 48 months
OS Rates at 12 Months, 24 Months, 36 Months and 48 Months in the FAS | 12, 24, 36 and 48 months
Investigator-assessed Time to Death or Distant Metastasis (TTDM) in the PPAS | From randomization until the first date of distant metastasis or death in the absence of distant metastasis (up to approximately 114 months)
Investigator-assessed TTDM in the FAS | From randomization until the first date of distant metastasis or death in the absence of distant metastasis (up to approximately 114 months)
Percentage of Participants With Adverse Events | Up to approximately 114 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (177):
- United States (25):
  - Stanford University, Palo Alto, California
  - Banner MD Anderson Cancer Center, Greeley, Colorado
  - Florida Cancer Specialists, Fort Myers, Florida
  - Cancer Care Centers of Brevard, Palm Bay, Florida
  - Woodlands Medical Specialists, P.A., Pensacola, Florida
  - Florida Cancer Specialist, North Region, St. Petersburg, Florida
  - Northwest Georgia Oncology Centers PC - Marietta, Marietta, Georgia
  - Illinois Cancer Care, Peoria, Illinois
  - New England Cancer Specialists, Brunswick, Maine
  - Southcoast Health System, Fairhaven, Massachusetts
  - Minnesota Oncology Hematology, Minneapolis, Minnesota
  - HCA Midwest Health, Kansas City, Missouri
  - Cox Health Systems, Springfield, Missouri
  - Optum Health Care, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Titan Health Partners LLC, d/b/a Astera Cancer Care, East Brunswick, New Jersey
  - San Juan Oncology Associates, Farmington, New Mexico
  - New York Oncology Hematology,P.C.-Albany, Albany, New York
  - Mount Sinai Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Prisma Health ? Upstate, Greenville, South Carolina
  - Tennessee Oncology Chattanooga, Chattanooga, Tennessee
  - Sarah Cannon Research Institute / Tennessee Oncology, Nashville, Tennessee
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
- Argentina (4):
  - CEMIC, Buenos Aires
  - Hospital Britanico de Buenos Aires, Ciudad Autonoma Buenos Aires
  - Clinica Universitaria Reina Fabiola, Córdoba
  - Sanatorio Parque S.A., Rosario
- Australia (6):
  - Blacktown Hospital, Blacktown, New South Wales
  - Macarthur Cancer Therapy Centre, Campbelltown, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Flinders Medical Centre, Bedford Park, South Australia
  - Monash Health Translational Precinct, Victoria, Victoria
  - Fiona Stanley Hospital, Bull Creek, Western Australia
- Austria (3):
  - Tiroler Landeskrankenanstalten Ges.M.B.H., Innsbruck
  - Kepler Universitätskliniken GmbH - Med Campus III, Linz
  - Klinik Penzing, Vienna
- Belgium (3):
  - GHdC Site Les Viviers, Charleroi
  - AZ Maria Middelares, Ghent
  - Jessa Zkh (Campus Virga Jesse), Hasselt
- Brazil (7):
  - Crio - Centro Regional Integrado de Oncologia, Fortaleza, Ceará
  - Centro Integrado de Oncologia de Curitiba, Curitiba, Paraná
  - Oncosite - Centro de Pesquisa Clinica Em Oncologia Ltda, Ijuí, Rio Grande do Sul
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
- Canada (5):
  - BC Cancer ? Abbotsford, Abbotsford, British Columbia
  - BC Cancer - Victoria, Victoria, British Columbia
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - William Osler Health System Brampton Civic Hospital, Brampton, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
- China (19):
  - Beijing Cancer Center, Beijing
  - Beijing Chest Hospital, Beijing
  - Xiangya Hospital Central South University, Changsha
  - Sichuan Provincial Cancer Hospital, Chengdu
  - Chongqing Cancer Hospital, Chongqing
  - Fujian Medical University Union Hospital, Fujian
  - Cancer Center, Sun Yat-sen University of Medical Sciences, Guangzhou
  - Hangzhou Cancer Hospital, Hangzhou
  - Shandong Cancer Hospital, Jinan
  - Zhongda Hospital Affiliated to Southeast University, Nanjing
  - The affiliated hospital of Qingdao university, Qingdao
  - Shanghai Chest Hospital, Shanghai
  - Cancer Hospital of Shantou University Medical College, Shantou
  - Shanxi Provincial Cancer Hospital, Taiyuan
  - Tianjin Cancer Hospital, Tianjin
  - The 2nd School of Medicine, WMU, Wenzhou
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou
  - Henan Cancer Hospital, Zhengzhou
- France (6):
  - CHU Angers, Angers
  - Centre Francois Baclesse, Caen
  - Hopital Nord AP-HM, Marseille
  - Clinique Clémentville, Montpellier
  - Hopital Robert Schuman, Vantoux
  - Institut Gustave Roussy, Villejuif
- Germany (4):
  - Klinikum Braunschweig, Braunschweig
  - Klinikum Koeln-Merheim, Cologne
  - Thoraxklinik Heidelberg gGmbH, Heidelberg
  - Universitätsklinikum Regensburg, Regensburg
- Greece (3):
  - General Hospital "G.Papanikolaou", Asvestochóri
  - Sotiria Hospital, Athens
  - Agioi Anargyroi Cancer Hospital, Kifissia
- Hong Kong (4):
  - Princess Margaret Hospital, Oncology, Hong Kong
  - Queen Elizabeth Hospital, Hong Kong
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong
  - Tuen Mun Hospital, Hong Kong
- Hungary (3):
  - Pécsi Tudományegyetem, Pécs
  - Szent Borbala Korhaz, Tatabánya
  - Tudogyogyintezet Torokbalint, Törökbálint
- Israel (4):
  - Soroka Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
- Italy (11):
  - Istituto Nazionale per lo Studio e la Cura dei Tumori Fondazione G. Pascale, Napoli, Campania
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola, Meldola, Emilia-Romagna
  - Azienda Ospedaliero Universitaria di Parma, Parma, Emilia-Romagna
  - Policlinico Universitario Campus Biomedico, Rome, Lazio
  - IRCCS Istituto Regina Elena (IFO), Rome, Lazio
  - IRCCS AOU San Martino - IST, Genoa, Liguria
  - A.O. Spedali Civili Di Brescia-P.O. Spedali Civili, Brescia, Lombardy
  - Azienda Socio Sanitaria Territoriale Niguarda (Ospedale Niguarda Ca' Granda), Milan, Lombardy
  - Fondazione IRCCS Policlinico San Matteo, Pavia, Lombardy
  - Azienda Ospedaliera Universitaria Pisana - Ospedale Cisanello, Pisa, Tuscany
  - Azienda ULSS 8 Berica, Vicenza, Veneto
- Japan (13):
  - Aichi Cancer Center, Aichi
  - National Cancer Center East, Chiba
  - National Hospital Organization Himeji Medical Center, Hyōgo
  - Kitasato University Hospital, Kanagawa
  - Kyoto University Hospital, Kyoto
  - Sendai Kousei Hospital, Miyagi
  - Niigata Cancer Center Hospital, Niigata
  - Kindai University Hospital, Osaka
  - Saitama Cancer Center, Saitama
  - Shizuoka Cancer Center, Shizuoka
  - National Cancer Center Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
  - Wakayama Medical University Hospital, Wakayama
- Netherlands (4):
  - Meander Medisch Centrum, Amersfoort
  - Amphia Ziekenhuis, Breda
  - Medisch Centrum Haaglanden, locatie Antoniushove, Leidschendam
  - Zuyderland Medisch Centrum - Sittard Geleen, Sittard-Geleen
- Auckland City Hospital, Cancer and Blood Research, Auckland, New Zealand
- Poland (5):
  - Uniwersyteckie Centrum Kliniczne, Gda?sk
  - Szpital Kliniczny MSWiA z Warmi?sko-Mazurskim Centrum Onkologii, Olsztyn
  - Mazowieckie Centrum Leczenia Chorob Pluc I Gruzlicy, Otwock
  - Narod.Inst.Onkol. im. M.Sklodowskiej - Curie-Panst.Inst.Bad, Warsaw
  - Dolnoslaskie Centrum Onkologii, Pulmonologii i Hematologii, Wroc?aw
- Portugal (4):
  - IPO de Coimbra, Coimbra
  - Hospital da Luz, Lisbon
  - Hospital CUF Porto, Porto
  - IPO do Porto, Porto
- South Korea (14):
  - Chungbuk National University Hospital, Cheongju-si
  - Kyungpook National University Chilgok Hospital, Daegu
  - National Cancer Center, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - St. Vincent's Hospital, Gyeonggi-do
  - Ajou University Medical Center, Gyeonggi-do
  - Pusan National University Yangsan Hospital, Gyeongsangnam-do
  - Gachon University Gil Medical Center, Incheon
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Ulsan University Hosiptal, Ulsan
- Spain (9):
  - Hospital Son Llatzer, Palma de Mallorca, Balearic Islands
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Provincial de Castellon, Castellon, Castellon
  - Complejo Hospitalario Universitario A Coruña (CHUAC), A Coruña
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario Carlos Haya, Málaga
  - Hospital Universitario Virgen del Rocio, Seville
- Taiwan (2):
  - China Medical University Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei
- Thailand (4):
  - Vajira Hospital, Bangkok
  - Rajavithi Hospital, Bangkok
  - Ramathibodi Hospital;Medicine/Oncology, Bangkok
  - Songklanagarind Hospital, Songkhla
- Turkey (Türkiye) (10):
  - Adana Baskent University Medical Faculty, Adana
  - Ankara University Medical Faculty, Ankara
  - Hacettepe Universitesi Tip Fakultesi Hastanesi, Ankara
  - Gazi University Medical Faculty, Oncology Hospital, Ankara
  - Ege University Medical Faculty, Bornova, ?zm?r
  - Dicle University Faculty of Medicine, Diyarbakır
  - Trakya Universitesi Tip Fakultesi, Medikal Onkoloji Bilim Dali, Balkan Yerleskesi, Edirne
  - Istanbul University Cerrahpasa Faculty of Medicine, Istanbul
  - Medipol University Medical Faculty, Istanbul
  - Inonu University Faculty of Medicine Turgut Ozal Medical Center, Malatya
- United Kingdom (4):
  - Birmingham Heartlands Hospital, Birmingham
  - Addenbrooke's NHS Trust, Cambridge
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Christie Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing